CLINICAL TRIAL: NCT01985841
Title: Phase II, Open-label Non-randomized Trial to Investigate the Efficacy of Bevacizumab in Combination With Dose Dense Sequential Chemotherapy in the Neo-adjuvant Setting for HER2 Negative Breast Cancer Patients
Brief Title: Bevacizumab in Combination With Chemotherapy in the Neo-adjuvant Setting for HER2 (-) Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/10.15
Record Dates: First submitted 2013-09-13; First posted 2013-11-15 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Primary operable breast cancer; HER2- negative; bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab/FEC/Docetaxel (Experimental): Bevacizumab plus 5-Fluorouracil/Epirubicin/Cyclophosphamide (FEC) -> Bevacizumab plus Docetaxel
  Interventions: Drug: Bevacizumb; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumb — Avastin
  Other Names: Bevacizumab: 10 mg/kg for up to 8 cycles from date of first dose; (cycle repeated every two weeks)
Drug: 5-Fluorouracil — 5-FU
  Other Names: 5-Fluorouracil: 700mg/m2 for up to 4 cycles from date of first dose; (cycle repeated every two weeks)
Drug: Epirubicin — Farmorubicin
  Other Names: Epirubicin: 75mg/m2 for up to 4 cycles from date of first dose; (cycle repeated every two weeks)
Drug: Cyclophosphamide — Endoxan
  Other Names: Cyclophosphamide: 700mg/m2 for up to 4 cycles from date of first dose; (cycle repeated every two weeks)
Drug: Docetaxel — Taxotere
  Other Names: Docetaxel: 75mg/m2 for up to 4 cycles from date of first dose; (cycle repeated every two weeks)

SUMMARY:
Investigators propose to study the efficacy of Bevacizumab plus systemic chemotherapy prior to surgery in order to make a locally advanced tumor operable. Treatment is thus expected to induce a maximum tumor shrinkage within a short period (usually 3-6 months). In addition Bevacizumab (Avastin) is to be administered as early as possible during the disease stages. The primary aim of this study is to evaluate the preliminary antitumor activity in terms of pathological complete responses (pCR) of bevacizumab in combination with chemotherapy.

DETAILED DESCRIPTION:
The aim of administering systemic therapy prior to surgery is to make a locally advanced tumor operable or to allow conservative surgery in the case of a T2-T3 tumor. Therefore, treatment is expected to induce a maximum tumor shrinkage within a short period. In addition and based on the anti-angiogenic MoA, bevacizumab (Avastin) is to be administered as early as possible during the disease stages. Bevacizumab has already been tested in the neoadjuvant setting with encouraging results. In a first trial patients with inoperable locally advanced breast cancer received docetaxel with or without bevacizumab with five clinical Complete Responses and 24 Partial Responses. In a second trial there was also reported the results of the combination of bevacizumab with doxorubicin and docetaxel for the treatment of inflammatory breast cancer. Then, a set of studies of primary therapy exploring the activity of different regimens have confirmed the role of baseline pathological features of the tumor in predicting the responsiveness to primary therapy. A 22% pathological complete responses (pCR) rate has been achieved in a study combining bevacizumab together with Xeloda and Taxotere suggesting that bevacizumab addition to chemotherapy in the neoadjuvant treatment is feasible showing promising activity while no unexpected toxicities were reported.

Thus, a very high interest exists from our clinicians mostly within our cooperative groups which cover the largest national oncology centers to be involved and run such a study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologic proven, corebiopsied, invasive ductal adenocarcinoma of the breast >2 cm in size and of any N stage (clinical and/or radiological T-stage > T1, including T4d), scheduled to receive preoperative chemotherapy.
* Age 18-70 years
* ECOG performance-status ≤1
* No prior or current neoplasm except for curatively treated non melanoma skin cancer, in situ carcinoma of the cervix
* No distant disease/secondary carcinoma
* Normal cardiac function
* Results of the following assessments at the time of inclusion must be available:

  1. bilateral Mammography (before enrolment)
  2. histology
  3. grading
  4. hormone-receptor-status
  5. HER2 status negative (is defined as FISH/CISH negative or IHC0 or IHC1+, or IHC2+ and FISH/CISH negative)
* Laboratory requirements (within 1 week before enrolment):

  1. Hematology: Neutrophils ≥ 1.5 x 109/l, Platelets ≥ 100 x 109/l, Hemoglobin>11 g/dl
  2. Hepatic function: Total bilirubin < 1 x ULN, SGOT and SGPT < 1.5 x ULN, Alkaline phosphatases < 1.5 x ULN. In case of abnormal values, the liver function tests have to be repeated within 3 days before study treatment.
  3. Renal function: Creatinine < 1 x ULN
  4. Urinalysis: Urine dipstick of proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1 g of protein / 24 hours.
* Signed and dated Informed Consent before the start of specific protocol procedures
* If of childbearing potential, negative pregnancy test

Exclusion Criteria:

* Cytological only confirmation of diagnosis
* Lobular or other non-ductal types of breast cancer
* Pregnant, or lactating patients; patients of childbearing potential must implement adequate contraceptive measures during study participation
* Pre-existing motor or sensory neurotoxicity of a severity > grade 2 by NCI-CTC AE
* Preoperative local treatment for breast cancer (i.e. incomplete surgery, radiotherapy)
* Prior or concurrent systemic antitumor therapy
* Evidence of wound healing complications, bone fracture, ulcer or the presence of clinically significant peripheral vascular disease
* Clinically significant cardiac disease e.g. congestive heart failure.
* Other serious illness or medical condition-uncontrolled hypertension or high risk uncontrolled arrythmias -history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent-active uncontrolled infection-unstable peptic ulcer, unstable diabetes mellitus or other contraindication for the use of corticosteroids
* Known hypersensitivity reaction to the compounds or incorporated substances.
* Evidence of bleeding diathesis or coagulopathy
* The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR, or appropriate monitoring test is within therapeutic limits and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of randomization. Patients not receiving anti coagulant medication must have an INR ≤ 1.5 an aPTT ≤ 1.5 x ULN within 7 days of randomization.
* Ongoing treatment with aspirin (> 325mg / day) or other medications known to predispose to gastrointestinal ulceration.
* Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrolment.
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
* Treatment with an investigational drug within 30 days prior to study entry.
* Legally incapacitated and/or other circumstances which make it undesirable for the subject to understand the nature, meaning and consequences of the clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Complete Response | On week 8 and 16
  Patients will be assessed for tumor response on week 8 and on week 16. Patients with tumor reduction will proceed on surgery. Histology report will confirm the complete or partial responses to chemotherapy.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Patients overall survival will be calculated from the date of the first chemotherapy cycle until the date of death from any cause
Progression Free Survival | 5 years
  Patients will be assessed every 8 weeks, from date of randomization until the end of treatment and then every 3 months until the date of first documented disease progression or date of death from any cause, whichever came first, up to 260 weeks (65 months).

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavroudis, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (6):
- Greece (6):
  - "IASO" General Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Euromedica" Hospital of Thessaloniki, Thessaloniki
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki